CLINICAL TRIAL: NCT01767779
Title: Potential EEG Biomarkers and Antiepileptogenic Strategies for Epilepsy in TSC
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); The University of Texas Health Science Center, Houston (Other); University of California, Los Angeles (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Martina Bebin, Associate Professor of Neurology, University of Alabama at Birmingham
Other Study IDs: 1P20NS080199-01 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Epilepsy; TSC; Tuberous Sclerosis Complex; Infants; Seizures; Biomarkers; EEG
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single venous blood sample will be drawn from the child and parents/family guardian for future research studies and future genetic testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- seizure free infants with dx of TSC: infants that are seizure free at the time of the study enrollment and meets genetic or clinical diagnostic criteria for TSC
- Parents or family guardian of cohort 1: Parent or family guardian of infants that are seizure free at the time of the study enrollment and meets genetic or clinical diagnostic criteria for TSC.

SUMMARY:
To determine whether EEGs during infancy is a reliable biomarker to identify TSC patients that will develop infantile spasms/epilepsy in the near future and thus are appropriate candidates for an antiepileptogenic drug trial. Since not all patients with TSC develop epilepsy, it would be useful to have a biomarker that could predict those patients destined to have epilepsy and thus identify those TSC patients most appropriate for an antiepileptogenic drug trial. A recent study suggests that treating TSC patients with an abnormal EEG prior to onset of infantile spasms with vigabatrin may improve neurological outcome, but the use of EEG as a reliable biomarker of future epilepsy has not been rigorously validated. In this specific aim, we will test the reliability of EEG in predicting future development of infantile spasms or epilepsy in TSC patients during the first year of life.

DETAILED DESCRIPTION:
Current therapeutic approaches for epilepsy primarily represent symptomatic treatments that suppress seizures, but have not been demonstrated to prevent epilepsy or modify disease progression. In recent years, there have been tremendous interest and effort by basic scientists and clinicians in epilepsy in developing disease-modifying or "antiepileptogenic" therapies. However, these efforts are hindered by a couple significant limitations: 1) difficulty in identifying an appropriate high-risk patient population in which a preventative approach is feasible and justifiable, and 2) lack of appropriate drug targets with antiepileptogenic properties. Tuberous Sclerosis Complex (TSC) is one of the most common genetic causes of epilepsy and a subset of TSC patients may represent a rational, feasible population to target with an antiepileptogenic approach for several reasons. First of all, some patients are diagnosed with TSC at a young age before the onset of epilepsy due to non-neurological findings - thus, it is feasible to identify these patients and initiate a potential antiepileptogenic treatment at an early stage of epileptogenesis. Second, these patients are at high risk for developing epilepsy (~80%) in the future, including infantile spasms (~35%), a particularly devastating type of childhood epilepsy with a poor prognosis - thus, initiating a therapy with potential side effects in a pre-symptomatic stage can likely be justified in TSC patients. Finally, the identification of the mTOR pathway in the pathophysiology of TSC suggests that mTOR inhibitors could have antiepileptogenic properties in TSC, as already supported by pre-clinical animal studies - thus, a rational mechanistically-based treatment potentially already exists and can be readily tested in TSC patients. However, there may be significant risks and side effects of mTOR inhibitors, especially during early childhood, such as chronic immunosuppression and theoretical effects on learning, growth, and development. Thus, before initiating an antiepileptogenic drug trial in TSC patients, it would be beneficial to obtain further evidence to optimize the selection criteria and treatment paradigms to maximize efficacy and minimize side effects of mTOR inhibitors.

The aim of this clinical trial is to determine whether EEGs during infancy is a reliable biomarker to identify TSC patients that will develop infantile spasms/epilepsy in the near future and thus are appropriate candidates for an antiepileptogenic drug trial.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* < 6 months of age; Seizure free at the time of study enrollment; and meets genetic or clinical diagnostic criteria for TSC (Tuberous Sclerosis), the latter based on current recommendations for diagnostic evaluation, such as physical exam, neuroimaging, echocardiogram.

Cohort 2

* Parent or family guardian of infant

Exclusion Criteria:

Cohort 1

* ≥ 6months of age; history of seizures and/or infantile spasms; patients receiving vigabatrin or any anti-epileptic medication or mTOR inhibitor prior to study enrollment Cohort 2
* not parent or family guardian

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants that are seizure free at the time of the study enrollment and meets genetic or clinical diagnostic criteria for TSC (determined as standard of care); parent/family guardian health status is unknown
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Identification of EEG biomarkers as predictors of developing epilepsy in infants with Tuberous Sclerosis Complex | 3 years
  Physical/neurological exam, Video EEG, Developmental assessments, Blood draw from child and parents/guardian, and Seizure diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Bebin, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas in Houston, Houston, Texas